CLINICAL TRIAL: NCT01346137
Title: An Exploratory Study of a COX-2 Inhibitor(Meloxicam) for Prevention of Ovulation
Brief Title: Study of a COX-2 Inhibitor for Prevention of Ovulation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Chileno de Medicina Reproductiva (Other)
Collaborators: CONRAD (Other)
Responsible Party: Cristián Jesam Gaete, ICMER
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIG-10-131
Record Dates: First submitted 2011-04-19; First posted 2011-05-02 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-03

CONDITIONS: Rupture; Graafian Follicle
Keywords: ovulation; unruptured luteinized follicle; meloxicam
MeSH Terms: conditions — Rupture | interventions — Meloxicam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- meloxicam (Experimental): 15 mg versus 30 mg per day P.O for 15 days, during 3 menstrual cycles
  Interventions: Drug: Meloxicam

INTERVENTIONS:
Drug: Meloxicam — 15 mg versus 30 mg per day P.O. for 15 days during 3 menstrual cycles

SUMMARY:
In this study the investigators propose to evaluate a COX-2 inhibitor(meloxicam) to assess its effect on follicular development and find out if this regimen delays or blocks ovulation while maintaining ovarian cyclicity. The investigators intend to administer 15 mg or 30 mg of meloxicam per day for 18 days starting on day 5 after onset of menses during 3 continuous cycles. The 3 treatment cycles will be preceded and followed by control cycles with no treatment. Ovulation or lack there of will be monitored by transvaginal ultrasound examinations (TVUs), estradiol, luteinizing hormone (LH), and progesterone levels in multiple blood samples in each cycle. The investigators will recruit a total of 56 women. Each woman will be randomly assigned to 1 of the 2 dose regimens of meloxicam, with 28 women assigned to each of the 2 dose regimens. Participating women will demonstrate an ovulatory cycle before starting meloxicam treatment and will be protected from pregnancy by prior sterilization.

DETAILED DESCRIPTION:
In a recent study, following follicular development by daily ultrasound examinations in 22 women, meloxicam was administered when the dominant follicle reached a diameter of 18 mm (Jesam, Salvatierra et al. 2010). Results from this study indicate that meloxicam 30 mg given for five days in late follicular phase was more effective at delaying follicular rupture than 15 mg. Follicular rupture was delayed more than 48 hours in 11/22 (50%) volunteers in the group treated with 15 mg/day and in 20/22 (91%) volunteers in the group treated with 30 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Proven fertility in the past
* 18- 40 years old
* Regular menstrual cycles in the past 3 months (24-35 days)
* Surgically sterilized
* Non-lactating
* Hemoglobin of at least 11 g/dl
* Willing to give informed consent in writing

Exclusion Criteria:

* Allergy to meloxicam, aspirin, or other NSAIDs
* Currently pregnant or breast feeding
* History of gastrointestinal problems like stomach ulcer, bleeding or bowel problems
* History of heart attack, stroke, or blood clot
* Hemorrhagic or coagulation disorders
* Known liver and renal disorder
* History of or signs and symptoms of cancer, hyperprolactinemia, bloody breast discharge, diabetes, or any endocrine disturbance
* History of asthma, skin or mucosal allergies
* Hypertension: systolic blood pressure > 135 mm Hg or diastolic blood pressure >85 mmHg
* History of mental illness including depression or epilepsy
* Cigarette smoker
* Habitual user of anti-inflammatory drugs
* Alcoholism or any drug abuse
* Use of anticoagulants or steroids

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Test the efficacy of meloxicam in preventing ovulation as measured by ovarian follicular development and delay in rupture when is administered daily for 18 days, starting on the 5th day of the cycle. | 3 menstrual cycles treated (3 months)
  To assess follicular outcomes transvaginal ultrasound will be done to all participants during treatment cycles

SECONDARY OUTCOMES:
Occurrence of functioning corpus luteum subsequent to unruptured follicles | 3 menstrual cycles treated (3 months)
Bleeding pattern during treatment with meloxicam | 3 menstrual cycles treated (3 months)
Incidence of adverse events | 3 menstrual cycles treated (3 months)
  In all cycles adverse events will be evaluated with a questionnaire performed in all visits
Pharmacokinetics of meloxicam | 1 menstrual cycle (1 month)
  During the first treatment cycle, plasma levels of meloxicam will be measured in all participants to evaluate levels obtained with the administration of the drug for 15 consecutive days. Levels of the drug will be correlate with follicular outcomes
Levels of estradiol | 3 menstrual cycles treated (3 months)
Levels of progesterone | 3 menstrual cycles (3 months)
Levels of LH | 3 menstrual cycles (3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Cristián Jesam, MD, Principal Investigator — Instituto Chileno de Medicina Reproductiva
Locations (1):
- Instituto Chileno de Medicina Reproductiva (ICMER), Santiago, Chile

REFERENCES:
- [Background] Jesam C, Salvatierra AM, Schwartz JL, Croxatto HB. Suppression of follicular rupture with meloxicam, a cyclooxygenase-2 inhibitor: potential for emergency contraception. Hum Reprod. 2010 Feb;25(2):368-73. doi: 10.1093/humrep/dep392. Epub 2009 Nov 19. PMID 19933235
- [Background] Bata MS, Al-Ramahi M, Salhab AS, Gharaibeh MN, Schwartz J. Delay of ovulation by meloxicam in healthy cycling volunteers: A placebo-controlled, double-blind, crossover study. J Clin Pharmacol. 2006 Aug;46(8):925-32. doi: 10.1177/0091270006289483. PMID 16855077
- [Derived] Jesam C, Salvatierra AM, Schwartz JL, Fuentes A, Croxatto HB. Effect of oral administration of a continuous 18 day regimen of meloxicam on ovulation: experience of a randomized controlled trial. Contraception. 2014 Aug;90(2):168-73. doi: 10.1016/j.contraception.2014.04.011. Epub 2014 May 5. PMID 24909636
- See also: Related Info — http://www.icmer.org